CLINICAL TRIAL: NCT06451770
Title: A Phase 1b Single Ascending Dose Study to Evaluate the Safety of VERVE-201 in Patients With Refractory Hyperlipidemia
Brief Title: Phase 1b Study of VERVE-201 in Patients With Refractory Hyperlipidemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Verve Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VT-20101
Record Dates: First submitted 2024-06-04; First posted 2024-06-11 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Hypercholesterolemia; Hypertriglyceridemia; Refractory Hyperlipidemia
Keywords: VERVE-201; Gene Editing; Base Editing; Refractory Hypercholesterolemia; ANGPTL3; ASCVD; Refractory Hypertriglyceridemia; Refractory Hyperlipidemia; Familial Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia; Hypertriglyceridemia; Hyperlipidemias; Hyperlipoproteinemia Type II

STUDY DESIGN:
Intervention Model Description: Single ascending dose escalation/adaptive design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Cohort 1: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-201.
  Interventions: Drug: VERVE-201
- Cohort 2: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-201.
  Interventions: Drug: VERVE-201
- Cohort 3: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-201.
  Interventions: Drug: VERVE-201
- Cohort 4: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-201.
  Interventions: Drug: VERVE-201
- Cohort 5: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-201.
  Interventions: Drug: VERVE-201
- Cohort 6: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-201.
  Interventions: Drug: VERVE-201

INTERVENTIONS:
Drug: VERVE-201 — Intravenous (IV) infusion

SUMMARY:
VT-20101 is an Open-label, Phase 1b, Single-ascending dose study that will evaluate the safety of VERVE-201 administered to patients with Refractory Hyperlipidemia.

VERVE-201 uses base-editing technology designed to inactivate the expression of the ANGPTL3 gene in the liver and lower circulating low-density lipoprotein cholesterol (LDL-C) and triglycerides. This study is designed to determine the safety and pharmacodynamic profile of VERVE-201 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Refractory hypercholesterolemia
* Refractory hypertriglyceridemia

Exclusion Criteria:

* Active or history of chronic liver disease
* Current treatment with monoclonal antibody targeting ANGPTL3 or prior treatment within specified timeframe
* Clinically significant or abnormal laboratory values as defined by the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Up to Day 365

SECONDARY OUTCOMES:
Evaluation of maximum observed concentration (Cmax) | Up to Day 365
Evaluation of time to maximum observed concentration (tmax) | Up to Day 365
Evaluation of terminal elimination half-life (t1/2) | Up to Day 365
Percent and absolute change from baseline in serum ANGPTL3 concentration | Up to Day 365
Percent and absolute change from baseline in serum LDL-C | Up to Day 365
Percent and absolute change from baseline in serum triglycerides | Up to Day 365

CONTACTS AND LOCATIONS:
Locations (10):
- Australia (2):
  - Clinical Study Center, Adelaide
  - Clinical Study Center, Melbourne
- Canada (3):
  - Clinical Study Center, Chicoutimi
  - Clinical Study Center, Montreal
  - Clinical Study Center, Toronto
- South Africa (2):
  - Clinical Study Center, Cape Town
  - Clinical Study Center, Johannesburg
- United Kingdom (3):
  - Clinical Study Center, Liverpool
  - Clinical Study Center, London
  - Clinical Study Center, Manchester